CLINICAL TRIAL: NCT00743899
Title: Conservative Versus Aggressive Revascularization in Patients With Intermediate Lesions Undergoing Percutaneous Coronary Intervention With Angiography Guidance Alone (SMART-CASE)
Brief Title: Conservative Versus Aggressive Revascularization in Patients With Intermediate Lesions Undergoing Percutaneous Coronary Intervention With Angiography Guidance Alone
Acronym: SMART-CASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-06-027
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease
Keywords: Angioplasty, Transluminal, Percutaneous Coronary; Everolimus-eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The aggressive group
  Interventions: Procedure: The aggressive group
- 2 (Experimental): The conservative group
  Interventions: Procedure: The conservative group

INTERVENTIONS:
Procedure: The aggressive group — Stents were implanted in lesions with diameter stenosis >50% and RD ≥2.25 mm and balloon angioplasty was performed in lesions with diameter stenosis >50% and RD ≥2.0 mm and <2.25 mm.
  Arms: 1
Procedure: The conservative group — Stenting was performed only in lesions with diameter stenosis >70% and reference diameter (RD) ≥2.25 mm
  Arms: 2

SUMMARY:
The aim of this study was to compare conservative versus aggressive strategy in patients with intermediate lesions with angiography guidance alone.

DETAILED DESCRIPTION:
To investigate whether conservative revascularization using criteria of 70% diameter stenosis would be non-inferior to aggressive revascularization using criteria of 50% diameter stenosis in coronary intermediate lesions, we conducted the Conservative Revascularization versus Aggressive Revascularization for Coronary Stenting with Everolimus-Eluting Stents (SMART-CASE) trial.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate coronary lesion(s) (diameter stenosis between 50% and 70% by quantitative coronary analysis)
* Target lesion(s) must be located in a native coronary artery with diameter of ≥2.25 mm and ≤4.25 mm

Exclusion Criteria:

* cardiogenic shock
* myocardial infarction (MI) within 48 hours
* left main lesion
* drug-eluting stent implantation in the target vessel prior to enrollment
* ≥2 chronic total occlusions in major coronary territories
* history of bleeding diathesis or known coagulopathy
* gastrointestinal or genitourinary bleeding within 3 months or major surgery within 2 months
* platelet count <100,000 cells/mm3
* planned elective surgical procedure that would necessitate interruption of thienopyridine during the first 6 months after enrollment
* non-cardiac co-morbid conditions with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 899 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
A composite of all cause death, MI, or any revascularization | 1 year

SECONDARY OUTCOMES:
All cause Death | 1 years
Cardiac death | 1 years
Myocardial infarction (Q-wave and non-Q wave) | 1 years
Any revascularization | 1 years
Stent thrombosis | 1 years
Revascularization of target intermediate lesion | 1 years
Target vessel failure | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim J, Lim SH, Hahn JY, Jeong JO, Park YH, Chun WJ, Oh JH, Cho DK, Choi YJ, Im ES, Won KH, Lee SY, Kim SW, Choi KH, Lee JM, Park TK, Yang JH, Song YB, Choi SH, Gwon HC. Outcomes of Deferring Percutaneous Coronary Intervention Without Physiologic Assessment for Intermediate Coronary Lesions. Korean Circ J. 2025 Mar;55(3):185-195. doi: 10.4070/kcj.2023.0223. Epub 2024 Dec 2. PMID 39962964
- [Derived] Hahn JY, Choi SH, Jeong JO, Song YB, Choi JH, Park YH, Chun WJ, Oh JH, Cho DK, Lim SH, Choi YJ, Im ES, Won KH, Lee SY, Kim SW, Gwon HC. Conservative versus aggressive treatment strategy with angiographic guidance alone in patients with intermediate coronary lesions: The SMART-CASE randomized, non-inferiority trial. Int J Cardiol. 2017 Aug 1;240:114-119. doi: 10.1016/j.ijcard.2017.03.075. Epub 2017 Mar 18. PMID 28363687